CLINICAL TRIAL: NCT03837652
Title: Evaluation of Bone-borne Palatal Expander in Conjunction With Maxillary Osteotomy in the Treatment of Cleft Palate Patients
Brief Title: Bone-borne Palatal Expander With Corticotomy for Cleft Palate Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarah Ahmed Sameh (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sarah Ahmed Sameh, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SarahSamehMsc
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Cleft Palate
Keywords: Cleft palate; transverse discrepancy; palatal expansion; bone-borne
MeSH Terms: conditions — Cleft Palate | interventions — Maxillary Osteotomy

STUDY DESIGN:
Intervention Model Description: Before and after Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of bone-borne palatal expander & maxillary osteotomy — Application of bone-borne palatal expander in conjunction with maxillary osteotomy for expansion of constricted maxillae

SUMMARY:
The tooth-borne palatal expander has limitations in the subset of patients with scarred, constricted cleft palate. At times, although posterior expansion is successful, transverse expansion of the anterior palate (near the alveolar cleft) is inadequate.

Will the application of bone borne palatal expander combined with a corticotomy be more effective in the expansion of the constricted maxilla in cleft palate patients?

DETAILED DESCRIPTION:
Intervention:

Application of bone-borne palatal expander in conjunction with maxillary osteotomy for expansion of constricted maxillae for previously treated cleft palate patients.

o Preoperative Preparations: All data of the patient will be gathered including personal data, medical history, family history, and classification of palatal cleft will be registered;

* Laboratory investigations will be conducted (CBC, coagulation profile, weight). -Models from dental impressions are made to make standardized measurements which include:-
* IMD: distance between two lingual grooves of two opposing first molars
* ICD: distance between cusp tip if two opposing canines
* Alveolar cleft width
* Total palatal area
* The correct distractor module can be measured bone to bone with the fitting models to choose the distractor length.

  o General operative procedures
* The procedures will be performed under general anesthesia with nasotracheal intubation.
* Local anaesthesia with vasoconstriction Epinephrine 1:100:000 will be injected in the palatal mucosa and mucolabial fold.
* The palatal incision is done between the premolar and molar or between the premolars.
* Maxillary vestibular incision followed by lateral corticotomy.
* Placement of distractor plates horizontally and fixing it with self-drilling screws between two roots on each side.

  o Postoperative care:
* Cephalosporin antibiotic (Ceclor 125mg q12h) for 5 days.
* Otrivin nasal drops for 5 days.
* Pyrol drops Analgesic-Antipyretic Paracetamol (Acetaminophen )
* Patient will be followed up for 10 weeks.
* Activation of distractor is started after 1 week of surgery using the patient's key twice daily.
* Sample size Based on the previous paper by Carpenter et al. 2014, the expected difference in maximum expansion will be 7.3+/-5.4m. The investigators will need to study 6 patients to be able to reject the null hypothesis that this response difference is zero with probability (power) o.8. The type I error probability associated with this test of this null hypothesis is 0.05. This sample size is to be increased to 8 to compensate for possible losses during follow up. Sample size was calculated using PS: Power and Sample Size software version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA.)
* Recruitment Strategy
* Patients will be selected from outpatient clinic of Department of Oral and Maxillofacial surgery - Cairo University.
* Screening of patients will continue until the target population is achieved.
* Identifying and recruiting potential subjects is achieved through patient database.

B) Data collection, management, and analysis

* Data collection methods

  1. Plans for assessment and collection of outcome

     1. Amount of bone expansion will be measured by collecting linear measurements from CBCT and dental models.
     2. Patient satisfaction will be measured using patient chart.
  2. Plans to promote participant retention and complete follow-up

     1. Telephone numbers of all patients included the study will be recorded as a part of the written consent.
     2. All patients will be given a phone call at the time of the predetermined follow-up dates.
* Data management All data will be entered electronically. Patients' files are to be stored in numerical order and stored in secure and accessible place. All data will be maintained in storage for 1 year after completion of the study.
* Statistical methods Data will be analyzed using IBM SPSS advanced statistics (statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between before and after treatment for normality distributed numeric variables will be done using the paired t-test while for non- normally distributed numeric variables will be done by Wilcoxon sign test. A p-value less than or equal to 0.05 will be considered statistically significant.

  1. Outcome:

     A suitable statistical test will be used to evaluate palatal expansion.
  2. Methods for any additional analysis:

No additional subgroup analysis.

C) Monitoring

* Data monitoring Data monitoring committee is independent from the supplying company of the palatal expander.
* Harms Patient will be closely monitored throughout the post operative period and any notices adverse effects will be managed as seen appropriate
* Auditing:

Auditing of the study design will be done by the research committee of the Department of Oral and Maxillofacial Surgery, Faculty of Oral and Dental Medicine, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-syndromic cleft palate.
* Patients with constricted maxilla after surgical treatment of cleft palate.
* Patients failed orthodontic expansion.
* Patients age between 8 and 18 years.

Exclusion Criteria:

* Patients with systemic disease or bleeding disorders.
* Patients with syndromic cleft palate.
* Patients failed with tooth borne expansion.
* Patients with fistula in cleft palate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adequate maxillary expansion | 10-12 weeks post operatively
  Dental casts before treatment & immediately after completion of expansion to determine transverse changes in maxillary arch width measured in millimeter at the following sites:
  Intermolar width Intercanine width Interarch width 6
  CBCT before operation & immediately after completion of consolidation period (10 weeks). Distances measured on the coronal images in millimeters before treatment & after the end of the consolidation period:
  NFW4 & NFW6: Nasal floor width at the area of first premolars & first molars, 5mm above the most inferior part of nasal floor
  PBW4 & PBW6 : Palatal bone width at the level of a line connecting palatal root apex of first premolars & first molars
  IRD4: distance between palatal root apex of right & left first premolars
  IRD6: distance between palatal root apex of right & left first molars

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sameh, BDS, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Figueiredo DS, Cardinal L, Bartolomeo FU, Palomo JM, Horta MC, Andrade I Jr, Oliveira DD. Effects of rapid maxillary expansion in cleft patients resulting from the use of two different expanders. Dental Press J Orthod. 2016 Nov-Dec;21(6):82-90. doi: 10.1590/2177-6709.2016-001.aop. PMID 27683832
- [Background] Marazita ML, Mooney MP. Current concepts in the embryology and genetics of cleft lip and cleft palate. Clin Plast Surg. 2004 Apr;31(2):125-40. doi: 10.1016/S0094-1298(03)00138-X. PMID 15145658
- [Background] Aziz SR, Tanchyk A. Surgically assisted palatal expansion with a bone-borne self-retaining palatal expander. J Oral Maxillofac Surg. 2008 Sep;66(9):1788-93. doi: 10.1016/j.joms.2008.04.017. PMID 18718384
- [Background] Gunaseelan R, Cheung LK, Krishnaswamy R, Veerabahu M. Anterior maxillary distraction by tooth-borne palatal distractor. J Oral Maxillofac Surg. 2007 May;65(5):1044-9. doi: 10.1016/j.joms.2005.12.049. No abstract available. PMID 17448861
- [Background] Zandi M, Miresmaeili A, Heidari A. Short-term skeletal and dental changes following bone-borne versus tooth-borne surgically assisted rapid maxillary expansion: a randomized clinical trial study. J Craniomaxillofac Surg. 2014 Oct;42(7):1190-5. doi: 10.1016/j.jcms.2014.02.007. Epub 2014 Feb 22. PMID 24704281
- [Background] Lin L, Ahn HW, Kim SJ, Moon SC, Kim SH, Nelson G. Tooth-borne vs bone-borne rapid maxillary expanders in late adolescence. Angle Orthod. 2015 Mar;85(2):253-62. doi: 10.2319/030514-156.1. Epub 2014 Dec 9. PMID 25490552
- [Derived] Abouseada SAS, El-Ghafour MA, Kamel HM, Elbokle NN. Evaluation of transpalatal distraction in cleft palate patients. Oral Maxillofac Surg. 2024 Jun;28(2):967-974. doi: 10.1007/s10006-024-01207-4. Epub 2024 Jan 22. PMID 38253979